CLINICAL TRIAL: NCT06109311
Title: A Phase 3, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Once Daily Oral Orforglipron Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Insulin Glargine, With or Without Metformin and/or SGLT-2 Inhibitor
Brief Title: A Study of Orforglipron (LY3502970) in Participants With Type 2 Diabetes and Inadequate Glycemic Control With Insulin Glargine, With or Without Metformin and/or SGLT-2 Inhibitor
Acronym: ACHIEVE-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18567; J2A-MC-GZGW (Other: Eli Lilly and Company); U1111-1294-2797 (Other: UTN Number); 2023-507280-18-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the safety and efficacy of orforglipron. Participants will have Type 2 Diabetes (T2D) and have inadequate glycemic control with insulin glargine with or without metformin and/or SGLT-2 (sodium-glucose cotransporter-2) inhibitor. The study will last about 46 weeks and may include up to 20 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥7.0% [53 mmol/mol] to ≤10.5% [91 mmol/mol]
* Have been treated with stable doses of the same formulation of the following for ≥90 days prior to screening visit 1 and have maintained the same doses through randomization:

  * insulin glargine U-100 (100 U/mL) ≥0.25 U/kg/QD (units per kilogram per day) or ≥20 U/QD alone, or
  * insulin glargine U-100 (100 U/mL) ≥0.25 U/kg/QD or ≥20 U/QD in combination with
  * metformin, or
  * SGLT-2 inhibitor, or
  * both metformin and SGLT-2 inhibitor.
* Are of stable body weight (±5%) for at least 90 days prior to screening visit 1 and agree to not initiate an intensive diet or exercise program during the study with the intent of reducing body weight, other than the lifestyle and/or dietary measures for diabetes treatment.
* Have a Body Mass Index (BMI) ≥23.0 kg/m^2 at baseline.

Exclusion Criteria:

* Have New York Heart Association functional classification III-IV congestive heart failure.
* Have had any of the following cardiovascular conditions within 60 days prior to baseline.

  * acute myocardial infarction
  * cerebrovascular accident (stroke), or
  * hospitalization for congestive heart failure.
* Have acute or chronic hepatitis, including a history of autoimmune hepatitis, signs or symptoms of any other liver disease other than nonalcoholic fatty liver disease
* Have had chronic or acute pancreatitis any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Orforglipron Dose 1, 2: Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Orforglipron Dose 3: Change from Baseline in HbA1c | Baseline, Week 40
Percentage of Participants Who Achieved HbA1c <7.0% (53 millimoles per mole (mmol/mol)) | Baseline to Week 40
Percentage of Participants Who Achieved HbA1c ≤6.5% (48 mmol/mol) | Baseline to Week 40
Change from Baseline in Fasting Serum Glucose | Baseline, Week 40
Percentage Change from Baseline in Body Weight | Baseline, Week 40
Change from Baseline in Body Weight | Baseline, Week 40
Percentage Change from Baseline in non-HDL (non-high-density lipoprotein) Cholesterol | Baseline, Week 40
Percentage Change from Baseline in Triglycerides | Baseline, Week 40
Change from Baseline in Systolic Blood Pressure | Baseline, Week 40
Change from Baseline in Daily Insulin Glargine Dose | Baseline, Week 40
Percentage of Participants Who Achieved Weight Loss of ≥5% | Baseline to Week 40
Percentage of Participants Who Achieved Weight Loss of ≥10% | Baseline to Week 40
Percentage of Participants Who Achieved Weight Loss of ≥15% from Baseline | Baseline to Week 40
Change from Baseline in Short Form 36-Version 2 (SF-36v2) Acute Form Domain and Summary Scores | Baseline, Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (25):
  - MD First Research - Chandler, Chandler, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - SanRo Clinical Research Group, Bryant, Arkansas
  - Velocity Clinical Research, Gardena, Gardena, California
  - Loma Linda University Health System, Loma Linda, California
  - Western University of Health Sciences, Pomona, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Care Access - Brandon, Brandon, Florida
  - Encore Medical Research, Hollywood, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Orita Clinical Research, Decatur, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - St. Luke's Humphreys Diabetes Center: Boise, Boise, Idaho
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - The Research Group of Lexington, Lexington, Kentucky
  - Clinvest Headlands Llc, Springfield, Missouri
  - Richmond University Medical Center, Staten Island, New York
  - Velocity Clinical Research, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Lifedoc Research - Lenox Park Drive, Memphis, Tennessee
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
- Brazil (9):
  - CEDOES, Vitória, Espírito Santo
  - L2IP - Instituto de Pesquisas Clínicas, Brasília, Federal District
  - Quanta Diagnóstico e Terapia, Curitiba, Paraná
  - Insight Centro de Pesquisas, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
- China (10):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
- Japan (14):
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - MinamiAkatsukaClinic, Mito, Ibaraki
  - Matoba Internal Medicine Clinic, Ebina, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - Tama Center Clinic Mirai, Tama, Tokyo
  - Jinnouchi Hospital, Kumamoto
  - Kansai Electric Power Hospital, Osaka
  - Abe Clinic, Ōita
- Puerto Rico (2):
  - Centro de Endocrinologia y Nutricion, Caguas
  - FDI Clinical Research, San Juan
- Romania (10):
  - Diabdana, Oradea, Bihor County
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Geea Medical Easy Diet, Bucharest, București
  - Centrul Medical NutriLife, Bucharest, București
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest, București
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş, Mureș County
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Clinica Korall, Satu Mare

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) in Participants With Type 2 Diabetes and Inadequate Glycemic Control With Insulin Glargine, With or Without Metformin and/or SGLT-2 Inhibitor (ACHIEVE-5) — https://trials.lilly.com/en-US/trial/432400